CLINICAL TRIAL: NCT04808557
Title: SEM Evaluation of the Quantity of microRepair® Contained in Biorepair Total Protection Toothpaste Residue on Composite Surfaces of Orthodontic Buttons: an in Vivo Randomized Clinical Trial.
Brief Title: SEM Evaluation of the Quantity of microRepair® on Resin Composite Surfaces: an in Vivo Randomized Clinical Trial.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pavia (Other)
Responsible Party: Principal Investigator, Andrea Scribante, Research Resident, Principal Investigator, University of Pavia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2021-BUTTONS
Record Dates: First submitted 2021-03-16; First posted 2021-03-22 (Actual); Last update posted 2021-05-11 (Actual); Status verified 2021-05

CONDITIONS: Dental Caries; Dental Fillings
Keywords: Composite resins; Toothpastes; Orthodontic buttons
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Intervention Model Description: Volunteers will have buttons bonded on the vestibular surfaces of elements 1.4,1.5,1.6. Then, they will be randomly divided into two groups: Trial Group will use Biorepair Total Protection toothpaste for home oral care, whereas Control Group will use Sensodyne Repair & Protect for home oral care.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Trial Group (Active Comparator): Volunteers from this group will have bonded buttons on vestibular surfaces of elements 1.4, 1.5 and 1.6. Then they will use Biorepair Total Protection for home oral care for 30 days. In this time period, the buttons will be respectively debonded at 7 (1.4), 15 (1.5) and 30 (1.6) days after the bonding procedures, in order to be evaluated at SEM.
  Interventions: Other: Biorepair Total Protection
- Control Group (Active Comparator): Volunteers from this group will have bonded buttons on vestibular surfaces of elements 1.4, 1.5 and 1.6. Then they will use Sensodyne Repair & Protect for home oral care for 30 days. In this time period, the buttons will be respectively debonded at 7 (1.4), 15 (1.5) and 30 (1.6) days after the bonding procedures, in order to be evaluated at SEM.
  Interventions: Other: Sensodyne Repair & Protect

INTERVENTIONS:
Other: Biorepair Total Protection — Volunteers will use Biorepair Total Protection for home oral hygiene for the following 30 days from the bonding procedure.
  Arms: Trial Group
Other: Sensodyne Repair & Protect — Volunteers will use Sensodyne Repair & Protect for home oral hygiene for the following 30 days from the bonding procedure.
  Arms: Control Group

SUMMARY:
The aim of this study is to evaluate the quantity of Biorepair Total Protection toothpaste on composite surfaces inside oral cavity. Three orthodontic lingual buttons are bonded on the vestibular surfaces of upper right premolars (1.4 and 1.5) and upper right first molars (1.6) of volunteers. A composite resine is applied upon them. Then, after 7 days, 1.4 button will be debonded; after 15 days, 1.5 button are debonded; in the end, after 30 days the last button (1.6) is debonded. The buttons will be stored in sterile environment and then sent to laboratory for SEM evaluation.

DETAILED DESCRIPTION:
Orthodontic buttons are bonded on the vestibular surfaces of the upper right premolars (1.4 and 1.5) and the upper right first molar (1.6). A composite resin is polymerized on the top of the buttons. Then, participants are divided into two groups.

* Trial Group: participants from this group will receive a manual toothbrush and Biorepair Total Protection toothpaste for home oral hygiene after lunches.
* Control Groups: participants from this group will receive a manual toothbrush and Sensodyne Repair & Protect for home oral hygiene after lunches.

After 7 days from the procedure of bonding, the buttons on upper right first premolars (1.4) are debonded. After 15 days from the procedure of bonding, the buttons on upper right second premolars (1.5) are debonded. In the end, After 30 days from the procedure of bonding, the buttons on upper right first molars (1.6) are debonded.

Debonded buttons are then stored in sterile environment at 2-3°C temperature; successively, they are sent to laboratory for SEM evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients
* No current orthodontic treatment during the study
* No use of occlusal splint or retention device

Exclusion Criteria:

* Presence of white spot lesions on the vestibular surfaces of teeth
* Corrupted vestibular surfaces of teeth

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-03-24 (Actual); Primary Completion 2021-05-05 (Actual); Study Completion 2021-05-10 (Actual)

PRIMARY OUTCOMES:
% microRepair® on composite surfaces | 7 days from the bonding procedure.
  SEM evaluation of the percentage of microRepair® on composite surfaces.
% microRepair® on composite surfaces | 15 days from the bonding procedure.
  SEM evaluation of the percentage of microRepair® on composite surfaces.
% microRepair® on composite surfaces | 30 days from the bonding procedure.
  SEM evaluation of the percentage of microRepair® on composite surfaces.
Comparison with Control Group | 7 days from the bonding procedure.
  SEM evaluation of the possibile differences between Trial and Control Groups.
Comparison with Control Group | 15 days from the bonding procedure.
  SEM evaluation of the possibile differences between Trial and Control Groups.
Comparison with Control Group | 30 days from the bonding procedure.
  SEM evaluation of the possibile differences between Trial and Control Groups.

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Scribante, DDS, PhD., Principal Investigator — University of Pavia
Locations (1):
- Unit of Dental Hygiene - Section of Dentistry - Department of Clinical, Surgical, Diagnostic and Paediatrics - University of Pavia, Pavia, Lombardy, Italy

IPD SHARING:
Plan to Share IPD: No
Data will be available upon motivated request to Principal Investigator